CLINICAL TRIAL: NCT02357680
Title: Dagbøger Til Kritisk Syge Patienter Skrevet af pårørende: Betydning for Patient og pårørende Samt Effekt i Forhold Til Udvikling af Symptomer på Posttraumatisk Stress
Brief Title: Diaries for Critically Ill Patients Written by Relatives
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospitalsenheden Vest (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Principal Investigator, Anne Højager Nielsen, RN, MCN, ph.d. student, Hospitalsenheden Vest
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 45129
Record Dates: First submitted 2015-02-03; First posted 2015-02-06 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Stress Disorders, Post-Traumatic; Anxiety; Depression
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Relatives randomized to the intervention group is provied with a diary. Nurses advice relatives on how to write and use the diary under and after the patients stay in the ICU. A written description on how to use the diary is also provided.
  At least two photographs of the patient is taken by nurses. Photographs will first be included in the diary when full consent from the patient has been obtained.
  Patients and relatives recieve a questionaire 3 months after the patient has been dismissed from the ICU.
  Interventions: Other: Diary
- Control group (No Intervention): Standard Care. Patients and relatives recieve a questionaire 3 months after the patient has been dismissed from the ICU.

INTERVENTIONS:
Other: Diary — The intervention is a notebook in which the relative will be asked to keep a diary of the time when the patient is critically ill in the ICU. At least two photos of the patient will be added to the diary upon full consent from the patient.
  The diary contains a written description on how to use the diary during and after the patients stay in the ICU.
  Arms: Intervention group

SUMMARY:
This study will investigate the effect of diaries written by relatives for critically ill patients on the risk of posttraumatic stress symptoms.

Utilizing a randomized controlled design pairs of one patient and one relative will be assigned to either diary intervention or standard care. The effect of the diary will be evaluated using a questionnaire 3 months post charge.

The results of this study will add to the body of knowledge on how diaries may help critical care survivors and their relatives to proceed with their lives.

DETAILED DESCRIPTION:
Diaries written for critically ill patients has previously been shown to protect patient and relatives from new cases of post traumatic stress (Jones et al. 2010, Jones et al. 2012, Garrouste-Orgeas 2012). Furthermore it has been described how relatives and patients use diaries written by nurses to process the time they stayed in the intensive care unit (Egerod et al. 2011). This study will investigate if there is a similar effect, when relatives write the diary for the critically ill patient instead of nurses doing it as patients find it very valuable when relatives has contributed to the diary or when relatives presence has been documented in the diary (Engström et al. 2009).

The investigators hypothesis is that a diary written by relatives for critically ill patients will reduce the risk of developing symptoms of post traumatic stress in relatives and patients.

Design: randomized controlled study. Relative and patient are randomized as a pair to either intervention group (diary intervention) or control group (standard care). Relatives will be recruited to the study while the patient is critically ill in the ICU, the patient will be recruited when he or she is able to receive information about the study.

Intervention: Nurses guide the nearest relative (spouse, partner, child, parent or friend) to write a diary during the patients stay in the ICU and up to a month post discharge. The diary is a notebook which also contains a written instruction on how to write and use the diary during and after the time in the intensive care unit. At least two photographs of the patient is taken by the staff and added to the diary upon the patients consent.

Blinding: Due to the nature of the intervention neither caregivers nor participants can be blinded to the intervention. However, steps will be taken to ensure that the outcomes assessor is blinded.

Setting: the study will take place in the two ICUs (10 bed and 7 beds respectively) of the hospital unit Hospitalsenheden Vest, a 441 bed hospital serving 300.000 citizens. Both ICUs are mixed medical/surgical units.

Primary outcome: Risk of post traumatic stress symptoms (PTSS-14 (Twigg et al 2008).

Secondary outcomes: Anxiety and depressionsymptoms (HADS (Zigmond and Snaith 1983)) and general physical and psychological wellbeeing (SF-36 (Bjorner et al. 1998)).

Baseline data: To compare groups the following parameters will be recorded on all eligible patients. Patients: age, sex, education, marital status, diagnosis, SAPS-II score (Le Gall et al. 1993), hours on ventilator, LOS-ICU. Furthermore the following data will be recorded on participating relatives: age, sex, relation to patient, education and working status.

Sample size: Based on findings from a previous study (1) where the median PTSS-14 score was 24 (SD 12), alfa 5% and beta 80% and a minimal relevant difference of 4 points, 71 relative-patient pairs needs to be included in each group. To compensate for dropouts due to critical illness and death, 100 pairs will be included in each group. The data collection period is anticipated to last 24 months.

Follow-up: 3 months post ICU discharge all participants receive a questionnaire to be completed and returned by mail or email.

Statistical analysis will cover a comparison of mean and median values in the two study groups, supplemented by a stratified analysis to estimate risk reduction. Parametric and non-parametric test will be applied according to the nature of data.

Dissemination: Results, positive, negative or inconclusive will be published in an international peer-reviewed journal.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Expected to stay in ICU > 48 hours
* Expected to be on ventilator > 24 hours
* Has a close relative > 18 years old
* Speaking and understanding Danish.
* Expected to be able to deliver an informed consent later

Relative:

*Speaking and understanding Danish

Relative and patient are included in the study as a pair.

Exclusion Criteria:

* Patient staying less than 48 hours in ICU
* Patient less than 24 hours on ventilator
* Patient not able to give an informed consent to participate in study or patient dies in ICU (both relative and patient are excluded).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2015-03-15 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
PTSS-14 (Post Traumatic Stress Symptoms) | 3 months post discharge from ICU
  14 items inventory covering all symptoms of PTSD.

SECONDARY OUTCOMES:
HADS (Hospital Anxiety and Depression Scale) | 3 months post discharge from ICU
  14 items inventory assessing symptoms of anxiety and depression.
SF-36 | 3 months post discharge from ICU
  36 items inventory covering the general physical and psychological wellbeing of an individual.

CONTACTS AND LOCATIONS:
Overall Officials: Anne H Nielsen, RN, MCN, Principal Investigator — Hospitalsenheden Vest
Locations (2):
- Denmark (2):
  - Regionshospitalet Herning, Herning, Central Jutland
  - Regionshospitalet Holstebro, Holstebro, Central Jutland

REFERENCES:
- [Background] Jones C, Backman C, Capuzzo M, Egerod I, Flaatten H, Granja C, Rylander C, Griffiths RD; RACHEL group. Intensive care diaries reduce new onset post traumatic stress disorder following critical illness: a randomised, controlled trial. Crit Care. 2010;14(5):R168. doi: 10.1186/cc9260. Epub 2010 Sep 15. PMID 20843344
- [Background] Jones C, Backman C, Griffiths RD. Intensive care diaries and relatives' symptoms of posttraumatic stress disorder after critical illness: a pilot study. Am J Crit Care. 2012 May;21(3):172-6. doi: 10.4037/ajcc2012569. PMID 22549573
- [Background] Garrouste-Orgeas M, Coquet I, Perier A, Timsit JF, Pochard F, Lancrin F, Philippart F, Vesin A, Bruel C, Blel Y, Angeli S, Cousin N, Carlet J, Misset B. Impact of an intensive care unit diary on psychological distress in patients and relatives*. Crit Care Med. 2012 Jul;40(7):2033-40. doi: 10.1097/CCM.0b013e31824e1b43. PMID 22584757
- [Background] Egerod I, Christensen D, Schwartz-Nielsen KH, Agard AS. Constructing the illness narrative: a grounded theory exploring patients' and relatives' use of intensive care diaries. Crit Care Med. 2011 Aug;39(8):1922-8. doi: 10.1097/CCM.0b013e31821e89c8. PMID 21572330
- [Background] Engstrom A, Grip K, Hamren M. Experiences of intensive care unit diaries: 'touching a tender wound'. Nurs Crit Care. 2009 Mar-Apr;14(2):61-7. doi: 10.1111/j.1478-5153.2008.00312.x. PMID 19243522
- [Background] Twigg E, Humphris G, Jones C, Bramwell R, Griffiths RD. Use of a screening questionnaire for post-traumatic stress disorder (PTSD) on a sample of UK ICU patients. Acta Anaesthesiol Scand. 2008 Feb;52(2):202-8. doi: 10.1111/j.1399-6576.2007.01531.x. Epub 2007 Nov 14. PMID 18005373
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Bjorner JB, Kreiner S, Ware JE, Damsgaard MT, Bech P. Differential item functioning in the Danish translation of the SF-36. J Clin Epidemiol. 1998 Nov;51(11):1189-202. doi: 10.1016/s0895-4356(98)00111-5. PMID 9817137
- [Background] Le Gall JR, Lemeshow S, Saulnier F. A new Simplified Acute Physiology Score (SAPS II) based on a European/North American multicenter study. JAMA. 1993 Dec 22-29;270(24):2957-63. doi: 10.1001/jama.270.24.2957. PMID 8254858
- [Derived] Nielsen AH, Angel S, Egerod I, Hansen TB. The effect of diaries written by relatives for intensive care patients on posttraumatic stress (DRIP study): protocol for a randomized controlled trial and mixed methods study. BMC Nurs. 2018 Aug 16;17:37. doi: 10.1186/s12912-018-0306-y. eCollection 2018. PMID 30127664